CLINICAL TRIAL: NCT00160550
Title: A Double-blind, Multicenter, Randomized, Placebo-controlled Study to Evaluate the Efficacy and Safety of Adjunctive Treatment With 3000 mg/Day (Pediatric Target Dose of 60 mg/kg/Day) Oral Levetiracetam (LEV) (166, 250, and 500mg Tablets), in Adult and Pediatric Subjects (4-65 Years) Suffering From Idiopathic Generalized Epilepsy With Primary Generalized Tonic-clonic (PGTC) Seizures.
Brief Title: Study to Evaluate the Safety and Efficacy of Levetiracetam in Patients Suffering From Idiopathic Generalized Epilepsy With Primary Generalized Tonic-clonic Seizures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: N01057
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2009-09

CONDITIONS: Generalized Convulsive Epilepsy
Keywords: Idiopathic Generalized Epilepsy, tonic-clonic seizures; Levetiracetam, Keppra
MeSH Terms: conditions — Epilepsy, Generalized; Epilepsy, Idiopathic Generalized; Seizures | interventions — Levetiracetam

INTERVENTIONS:
Drug: Levetiracetam

SUMMARY:
This study will assess the efficacy, safety, and tolerability of adjunctive treatment with LEV (3,000 mg/day or a target dose of 60 mg/kg/day in children) compared to placebo in reducing PGTC seizures in subjects (4 - 65 years) suffering from idiopathic generalized epilepsy uncontrolled despite treatment with one or two concomitant AEDs.

ELIGIBILITY:
Inclusion Criteria:

* Subject with a confirmed diagnosis consistent with idiopathic generalized epilepsy experiencing primary generalized tonic-clonic seizures (IIE) that are classifiable according to the ILAE Classification of Epileptic Seizures.
* Presence of at least 3 PGTC seizures during the 8-week combined Baseline period.
* Absence of brain lesion documented on a CT scan or MRI.
* An EEG performed within 1 year of Visit 1 with features consistent with PGTC seizures or generalized idiopathic epilepsy.
* Male/female subject, >=4 or <=65 years of age at Visit 1.
* Subject on a stable dose of one or two AEDs during baseline.

Exclusion Criteria:

* Previous exposure to levetiracetam.
* History of partial seizures.
* History of convulsive or non-convulsive status epilepticus while taking concomitant AEDs within three months prior to Visit 1.

Ages: 4 Years to 65 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 154
Dates: Start 2001-09; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
The percentage reduction from the combined Baseline Period in the PGTC seizure frequency per week over the Treatment Period (up-titration + evaluation).

SECONDARY OUTCOMES:
Reduction during the Treatment Period in PGTC seizure frequency
Percentage reduction during the Treatment Period in seizure days
Responder rates in PGTC seizure frequency, and in seizure days of all types.
The safety parameters are the following: Laboratory tests; Adverse events; Electrocardiogram; Physical and neurological examinations

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — UCB Pharma

REFERENCES:
- [Result] Berkovic SF, Knowlton RC, Leroy RF, Schiemann J, Falter U; Levetiracetam N01057 Study Group. Placebo-controlled study of levetiracetam in idiopathic generalized epilepsy. Neurology. 2007 Oct 30;69(18):1751-60. doi: 10.1212/01.wnl.0000268699.34614.d3. Epub 2007 Jul 11. PMID 17625106
- [Result] Rosenfeld WE, Benbadis S, Edrich P, Tassinari CA, Hirsch E. Levetiracetam as add-on therapy for idiopathic generalized epilepsy syndromes with onset during adolescence: analysis of two randomized, double-blind, placebo-controlled studies. Epilepsy Res. 2009 Jul;85(1):72-80. doi: 10.1016/j.eplepsyres.2009.02.016. Epub 2009 Mar 26. PMID 19327967